CLINICAL TRIAL: NCT00362492
Title: 9-10 Days Versus Prolonged Thromboprophylaxis in Patients Without Evidence of Ultrasound Proximal Thromboembolism After Total Knee Joint Replacement: a Randomized Controlled Trial
Brief Title: Safety Study of Stopping Thromboprophylaxis Based on Ultrasound Results After Total Knee Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHRC-Prothege
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-10

CONDITIONS: Thromboembolism; Arthroplasty Replacement, Knee
Keywords: TKR; Ultrasonography; asymptomatic deep venous thrombosis; extended duration prophylaxis; short duration prophylaxis
MeSH Terms: conditions — Thromboembolism

INTERVENTIONS:
Procedure: Bilateral ultrasound examination 7+/- 2 after surgery

SUMMARY:
The purpose of this study is to determine whether stopping Low Molecular Weight Heparin (LMWH) thromboprophylaxis is safe after total knee joint replacement. The investigators select patients without proximal thromboembolism assessed by bilateral venous ultrasound examination 7-10 days after surgery. the investigators hypothesis is that stopping thromboprophylaxis is equally effective than prolonging thromboprophylaxis in order to prevent post-surgery complications in this population.

ELIGIBILITY:
Inclusion Criteria:

* First total knee joint replacement
* Signed informed consent

Non-inclusion Criteria:

* History of venous thromboembolism/major bleeding/Heparin induced thrombopenia
* Active cancer
* Long-term anticoagulation

Min Age: 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2004-06; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Thromboembolism occuring between day 7-35 ;
Major bleeding occuring between day 7-35 ;
LMWH induced thrombopenia
All cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Thérèse Barrellier, MD, Principal Investigator — Côte de Nacre University hospital; Claude Vielpeau, MD, Study Chair — Côte de Nacre University hospital
Locations (17):
- France (17):
  - Hospital Alençon, Alençon
  - Hospital University Angers, Angers
  - Clinique du Cèdre, Bois-Guillaume
  - Caen University hospital, Caen
  - Clinique St Marie, Chalon-sur-Saône
  - Hospital Val D'ariège, Foix
  - Hospital La Roche sur Yon, La Roche-sur-Yon
  - Mignot Hospital, Le Chesnay
  - Polyclinique de Riaumont, Liévin
  - Hospital University Lille, Lille
  - Hospital Nord Mayenne, Mayenne
  - Montluçon Hospital, Montluçon
  - Poitiers University Hospital, Poitiers
  - Reims University Hospital, Reims
  - Clinique St André, Reims
  - Clinique St Jean, Roubaix
  - Clinique St Jean Languedoc, Toulouse

REFERENCES:
- [Result] Barrellier MT, Lebel B, Parienti JJ, Mismetti P, Dutheil JJ, Vielpeau C; PROTHEGE study group; GETHCAM study group. Short versus extended thromboprophylaxis after total knee arthroplasty: a randomized comparison. Thromb Res. 2010 Oct;126(4):e298-304. doi: 10.1016/j.thromres.2010.07.018. Epub 2010 Aug 24. PMID 20797774